CLINICAL TRIAL: NCT01610791
Title: A Single Arm, Open Label Study to Assess the Safety, Tolerability and Efficacy of Tocilizumab in Active Rheumatoid Arthritis Patients With Inadequate Response to the DMARDs (REMISSION Study)
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to DMARDs (REMISSION)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22638
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks, total of 6 infusions

SUMMARY:
This open label, single arm study will assess the safety and efficacy of RoActemra/Actemra (tocilizumab) in patients with moderate to severe active rheumatoid arthritis who have an inadequate response to disease-modifying antirheumatic drugs (DMARDs). Patients will receive RoActemra/Actemra at a dose of 8 mg/kg intravenously every 4 weeks for 24 weeks (6 infusions).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe active rheumatoid arthritis (DAS28 > 3.2 at screening)
* Inadequate response to DMARDs
* Body weight < 150 kg

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months of enrollment
* Rheumatic autoimmune disease other than RA
* American College of Rheumatology (ACR) functional class IV
* Prior history of or current inflammatory joint disease other than RA
* Previous treatment with any biologic drug that is used in the treatment of RA
* Intraarticular or parenteral corticosteroids within 6 weeks prior to baseline
* Pregnant or lactating women
* Active current or history of recurrent infection, active TB within the previous 3 years, HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Morocco (8):
  - Casablanca
  - Fés
  - Kenitra
  - Khouribga
  - Marrakesh
  - Meknés
  - Rabat
  - Salé

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 milligrams per kilogram (mg/kg), intravenously (IV), once every 4 weeks for a total of 6 infusions.
Period: Overall Study
Arm/Group | Tocilizumab 8 mg/kg
Started | 121
Completed | 100
Not Completed | 21
Not completed — Lost to Follow-up | 7
Not completed — Adverse Event | 6
Not completed — Physician Decision | 1
Not completed — Adverse event and Investigator decision | 1
Not completed — Death | 1
Not completed — Not determined | 5

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population, defined as participants who received at least one dose of tocilizumab (baseline) and for whom data for at least one follow-up variable were available.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg, IV, once every 4 weeks for a total of 6 infusions.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 21

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With All-Cause Discontinuation of Tocilizumab by Study Visit
Description: Percentage of participants discontinuing study treatment for any reason at every visit; causes of discontinuation in the summary included AEs, deaths, lost to follo-wup, AE and investigator decision and 'not determined'.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: All enrolled participants were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 121
percentage of participants
  Week 4 | 3.3
  Week 8 | 3.3
  Week 12 | 2.5
  Week 16 | 2.5
  Week 20 | 2.5
  Week 24 | 3.3

2. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) to Highest Value
Description: The difference between baseline and highest values until Week 24 of ALT and AST. The values are measures as international units per liter (UI/L). The change was calculated as the value (highest) at a later timepoint up to Week 24, minus the value at Baseline.
Time Frame: Baseline through Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: UI/L
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 121
UI/L
  ALT | 23.6 (34.7)
  AST | 15.8 (22.1)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Difference in ALT from Baseline to Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Difference in AST from Baseline to Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change From Baseline Low-Density Lipoprotein (LDL) and Total Cholesterol (TC) to Highest Values
Description: Levels of LDL and TC were measured in milligrams/deciliter (mg/dL). Change in LDL and TC were calculated as the value (highest) through Week 24, minus the value at Baseline.
Time Frame: Baseline through Week 24
Population: Safety population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 120
mg/dL
  Total cholesterol | 57.2 (78.1)
  LDL cholesterol | 108.6 (106.2)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Diffrence in total cholesterol from baseline to Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Difference in LDL cholesterol from baseline to Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Percentage of Participants With Lipid Elevations by Study Visit
Description: Lipid panel assessed included TC, triglycerides, high-density lipoprotein (HDL), and LDL. Elevations were categorized as follows: LDL cholesterol: Optimal equals (=) less than (<)100 mg/dL, Near optimal=100-129 mg/dL, Borderline high 130-159 mg/dL, High 160-189 mg/dL, Very High ≥190 mg/dL; Total cholesterol: Desirable <200 mg/dL, Borderline high 200-239 mg/dL, High ≥240 mg/dL; HDL cholesterol: Low <40 mg/dL, High ≥60 mg/dL; Triglycerides: Normal <150 mg/dL, Borderline high 150-199 mg/dL, High 200-499 mg/dL, and Very high ≥500 mg/dL.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Safety population; n (number) = number of participants assessed for the parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 121
percentage of participants
  LDL Cholesterol: Optimal, Baseline (n=120) | 53.3
  LDL Cholesterol: Optimal, Week 4 (n=116) | 32.8
  LDL Cholesterol: Optimal, Week 8 (n=112) | 42.9
  LDL Cholesterol: Optimal, Week 12 (n=109) | 33.9
  LDL Cholesterol: Optimal, Week 16 (n=106) | 18.9
  LDL Cholesterol: Optimal, Week 20 (n=102) | 38.2
  LDL Cholesterol: Optimal, Week 24 (n=98) | 28.6
  LDL Cholesterol: Near Optimal, Baseline (n=120) | 30.8
  LDL Cholesterol: Near Optimal, Week 4 (n=116) | 31.9
  LDL Cholesterol: Near Optimal, Week 8 (n=112) | 22.3
  LDL Cholesterol: Near Optimal, Week 12 (n=109) | 25.7
  LDL Cholesterol: Near Optimal, Week 16 (n=106) | 17.9
  LDL Cholesterol: Near Optimal, Week 20 (n=102) | 22.5
  LDL Cholesterol: Near Optimal, Week 24 (n=98) | 27.6
  LDL Cholesterol: Borderline High, Baseline (n=120) | 12.5
  LDL Cholesterol: Borderline High, Week 4 (n=116) | 21.6
  LDL Cholesterol: Borderline High Week 8 (n=112) | 23.2
  LDL Cholesterol: Borderline High, Week 12 (n=109) | 20.2
  LDL Cholesterol: Borderline High, Week 16 (n=106) | 15.1
  LDL Cholesterol: Brderline High, Week 20 (n=102) | 25.5
  LDL Cholesterol: Borderline High, Week 24 (n=98) | 29.6
  LDL Cholesterol: High, Baseline (n=120) | 2.5
  LDL Cholesterol: High, Week 4 (n=116) | 7.8
  LDL Cholesterol: High, Week 8 (n=112) | 9.8
  LDL Cholesterol: High, Week 12 (n=109) | 14.7
  LDL Cholesterol: High, Week 16 (n=106) | 9.4
  LDL Cholesterol: High, Week 20 (n=102) | 10.8
  LDL Cholesterol: High, Week 24 (n=98) | 9.2
  LDL Cholesterol: Very High, Baseline (n=120) | 0.8
  LDL Cholesterol: Very High, Week 4 (n=116) | 6.0
  LDL Cholesterol: Very High, Week 8 (n=112) | 1.8
  LDL Cholesterol: Very High, Week 12 (n=109) | 5.5
  LDL Cholesterol: Very High, Week 16 (n=106) | 38.7
  LDL Cholesterol: Very High, Week 20 (n=102) | 2.9
  LDL Cholesterol: Very High, Week 24 (n=98) | 5.1
  TC: Desirable, Baseline (n=120) | 77.5
  TC: Desirable, Week 4 (n=116) | 58.6
  TC: Desirable, Week 8 (n=85) | 28.6
  TC: Desirable, Week 12 (n=109) | 56.0
  TC: Desirable, Week 16 (n=106) | 56.6
  TC: Desirable, Week 20 (n=103) | 52.4
  TC: Desirable, Week 24 (n=98) | 51.0
  TC: Borderline High, Baseline (n=120) | 18.3
  TC: Borderline High, Week 4 (n=116) | 25.0
  TC: Borderline High, Week 8 (n=85) | 28.6
  TC: Borderline High, Week 12 (n=109) | 23.9
  TC: Borderline High, Week 16 (n=106) | 26.4
  TC: Borderline High, Week 20 (n=103) | 28.2
  TC: Borderline High, Week 24 (n=98) | 26.5
  TC: High, Baseline (n=120) | 4.2
  TC: High, Week 4 (n=116) | 16.4
  TC: High, Week 8 (n=85) | 18.8
  TC: High, Week 12 (n=109) | 20.2
  TC: High, Week 16 (n=106) | 17.0
  TC: High, Week 20 (n=103) | 19.4
  TC: High, Week 24 (n=98) | 22.4
  HDL Cholesterol: Low, Baseline (n=49) | 28.1
  HDL Cholesterol: Low, Week 4 (n=47) | 12.9
  HDL Cholesterol: Low, Week 8 (n=54) | 17.7
  HDL Cholesterol: Low, Week 12 (n=42) | 11.0
  HDL Cholesterol: Low, Week 16 (n=51) | 24.5
  HDL Cholesterol: Low, Week 20 (n=52) | 22.3
  HDL Cholesterol: Low, Week 24 (n=48) | 19.4
  HDL Cholesterol: High, Baseline (n=49) | 12.4
  HDL Cholesterol: High, Week 4 (n=47) | 27.6
  HDL Cholesterol: High, Week 8 (n=54) | 30.1
  HDL Cholesterol: High, Week 12 (n=42) | 27.5
  HDL Cholesterol: High, Week 16 (n=51) | 23.6
  HDL Cholesterol: High, Week 20 (n=52) | 28.2
  HDL Cholesterol: High, Week 24 (n=48) | 29.6
  Triglycerides: Normal, Baseline (n=121) | 88.4
  Triglycerides: Normal, Week 4 (n=116) | 40.5
  Triglycerides: Normal, Week 8 (n=112) | 82.1
  Triglycerides: Normal, Week 12 (n=109) | 80.7
  Triglycerides: Normal, Week 16 (n=106) | 82.1
  Triglycerides: Normal, Week 20 (n=103) | 75.7
  Triglycerides: Normal, Week 24 (n=98) | 72.4
  Triglycerides: Borderline High, Baseline (n=121) | 8.3
  Triglycerides: Borderline High, Week 4 (n=116) | 28.4
  Triglycerides: Borderline High, Week 8 (n=112) | 8.0
  Triglycerides: Borderline High, Week 12 (n=109) | 8.3
  Triglycerides: Borderline High, Week 16 (n=106) | 8.5
  Triglycerides: Borderline High, Week 20 (n=103) | 9.7
  Triglycerides: Borderline High, Week 24 (n=98) | 16.3
  Triglycerides: High, Baseline (n=121) | 3.3
  Triglycerides: High, Week 4 (n=116) | 25.9
  Triglycerides: High, Week 8 (n=112) | 9.8
  Triglycerides: High, Week 12 (n=109) | 11
  Triglycerides: High, Week 16 (n=106) | 8.5
  Triglycerides: High, Week 20 (n=103) | 14.6
  Triglycerides: High, Week 24 (n=98) | 11.2
  Triglycerides: Very High, Baseline (n=121) | 0.0
  Triglycerides: Very High, Week 4 (n=116) | 5.2
  Triglycerides: Very High, Week 8 (n=112) | 0.0
  Triglycerides: Very High, Week 12 (n=109) | 0.0
  Triglycerides: Very High, Week 16 (n=106) | 0.9
  Triglycerides: Very High, Week 20 (n=103) | 0.0
  Triglycerides: Very High, Week 24 (n=98) | 0.0

5. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate (ESR; in millimeters per hour [mm/hour]) and global health assessment (participant-rated global assessment of disease activity using 10-mm visual analog assessment [VAS]); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 less than or equal to (≤3.2) = low disease activity, DAS28 greater than (>)3.2 to less than or equal to (≤) 5.1=moderate to high disease activity; DAS28 >5.1=high disease activity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
units on a scale
  Baseline (n=117) | 6.2 (1.5)
  Week 4 (n=116) | 4.0 (1.6)
  Week 8 (n=112) | 3.3 (1.4)
  Week 12 (n=109) | 2.8 (1.4)
  Week 16 (n=106) | 2.4 (1.4)
  Week 20 (n=103) | 2.1 (1.2)
  Week 24 (n=99) | 2.0 (1.3)

6. Secondary Outcome: Percentage of Participants by DAS28 Response Category
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 ≤3.2 =low disease activity, DAS28 >3.2 to ≤5.1=moderate to high disease activity; DAS28 >5.1=high disease activity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
percentage of participants
  DAS28 ≤3.2, Baseline (n=117) | 0.9
  DAS28 ≤3.2, Week 4 (n=116) | 31.9
  DAS28 ≤3.2, Week 8 (n=112) | 50.9
  DAS28 ≤3.2, Week 12 (n=109) | 67.9
  DAS28 ≤3.2, Week 16 (n=106) | 81.1
  DAS28 ≤3.2, Week 20 (n=103) | 88.3
  DAS28 ≤3.2, Week 24 (n=99) | 83.8
  DAS28 >3.2 and ≤5.1, Baseline (n=117) | 25.6
  DAS28 >3.2 and ≤5.1, Week 4 (n=116) | 43.1
  DAS28 >3.2 and ≤5.1, Week 8 (n=112) | 40.2
  DAS28 >3.2 and ≤5.1, Week 12 (n=109) | 25.7
  DAS28 >3.2 and ≤5.1, Week 16 (n=106) | 13.2
  DAS28 >3.2 and ≤5.1, Week 20 (n=103) | 9.7
  DAS28 >3.2 and ≤5.1, Week 24 (n=99) | 13.1
  DAS28 >5.1, Baseline (n=117) | 73.5
  DAS28 >5.1, Week 4 (n=116) | 25.0
  DAS28 >5.1, Week 8 (n=112) | 8.9
  DAS28 >5.1, Week 12 (n=109) | 6.4
  DAS28 >5.1, Week 16 (n=106) | 5.7
  DAS28 >5.1, Week 20 (n=103) | 1.9
  DAS28 >5.1, Week 24 (n=99) | 3.0

7. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement in Disease Activity
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. A reduction in DAS28 of at least 1.2 units was considered a clinically meaningful improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
percentage of participants
  Baseline | 0
  Week 4 | 76.7
  Week 8 | 91.1
  Week 12 | 91.7
  Week 16 | 96.2
  Week 20 | 98.1
  Week 24 | 100

8. Secondary Outcome: Time to Achieve Clinically Meaningful Reduction in DAS28
Description: A clinically meaningful improvement in DAS28 was defined as a reduction of at least 1.2 units. Time to achieving clinically meanigful improvement was calculated as the number of days from the first infusion to the first achievement of reduction of 1.2 units in DAS28.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
days | 44.7 (29.1)

9. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28 <2.6)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. Participants with a DAS28 score <2.6 were considered to have achieved remission.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
percentage of participants
  Baseline (n=117) | 0.0
  Week 4 (n=116) | 16.4
  Week 8 (n=112) | 30.4
  Week 12 (n=109) | 48.6
  Week 16 (n=106) | 63.2
  Week 20 (n=103) | 73.8
  Week 24 (n=99) | 74.7

10. Secondary Outcome: Percentage of Participants With a Response Assessed Using American College of Rheumatology (ACR) Criteria
Description: The ACR response rates ACR20, ACR50, ACR70 are defined as ≥20%, ≥50%, ≥70% improvement, respectively, in: swollen joint count (SJC) (66 joints) and tender joint count (TJC) (68 joints) and 3 of the following 5 assessments: Patient assessment of pain (VAS); Patient global assessment of disease activity (VAS); Investigator global assessment of disease activity (VAS); and acute phase response (ESR or CRP)
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 121
percentage of participants
  ACR20, Week 4 (n=121) | 62.0
  ACR20, Week 8 (n=112) | 73.2
  ACR20, Week 12 (n=109) | 78.9
  ACR20, Week 16 (n=106) | 85.8
  ACR20, Week 20 (n=103) | 90.3
  ACR20, Week 24 (n=99) | 87.9
  ACR50, Week 4 (n=116) | 27.6
  ACR50, Week 8 (n=112) | 50.0
  ACR50, Week 12 (n=109) | 63.3
  ACR50, Week 16 (n=106) | 77.4
  ACR50, Week 20 (n=103) | 85.4
  ACR50, Week 24 (n=99) | 80.8
  ACR70, Week 4 (n=115) | 6.9
  ACR70, Week 8 (n=112) | 29.5
  ACR70, Week 12 (n=109) | 32.1
  ACR70, Week 16 (n=106) | 48.1
  ACR70, Week 20 (n=103) | 56.3
  ACR70, Week 24 (n=99) | 61.6

11. Secondary Outcome: Swollen and Tender Joint Counts
Description: The following 28 joints were assessed by the physician for swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). The following 28 joints were assessed by the physician for tenderness : metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). The change in SJC and TJC was determined as the difference in values from baseline at each visit.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
joints
  SJC Baseline | 10.8 (7.4)
  SJC Week 4 | 4.8 (6.0)
  Change in SJC at Week 4 | 6.0 (6.5)
  SJC Week 8 | 3.1 (4.6)
  Change in SJC at Week 8 | 7.5 (6.8)
  SJC Week 12 | 2.8 (4.5)
  Change in SJC at Week 12 | 7.8 (6.9)
  SJC Week 16 | 1.8 (3.4)
  Change in SJC at Week 16 | 8.9 (7.4)
  SJC Week 20 | 0.9 (1.9)
  Change in SJC at Week 20 | 9.8 (7.4)
  SJC Week 24 | 1.0 (2.2)
  Change in SJC at Week 24 | 9.9 (7.6)
  TJC Baseline | 15.4 (8.8)
  TJC Week 4 | 9.3 (7.7)
  Change in TJC at Week 4 | 6.1 (7.6)
  TJC Week 8 | 6.2 (5.7)
  Change in TJC at Week 8 | 9.1 (7.2)
  TJC Week 12 | 4.7 (5.8)
  Change in TJC at Week 12 | 10.4 (7.4)
  TJC Week 16 | 3.3 (4.5)
  Change in TJC at Week 16 | 12.0 (7.6)
  TJC Week 20 | 2.5 (3.5)
  Change in TJC at Week 20 | 12.7 (7.8)
  TJC Week 24 | 2.3 (4.1)
  Change in TJC at Week 24 | 13.0 (8.4)

12. Secondary Outcome: Health Assessment Questionnaire (HAQ)
Description: HAQ was used to assess the physical ability and functional status of participants as well as quality of life. The disability dimension consists of 20 multiple-choice items concerning difficulty in performing 8 common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Participants choose from 4 response categories, ranging from 'without any difficulty' (Score=0) to 'unable to do' (Score=3). The change in HAQ was determined as the difference in values from baseline at each visit.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
score on a scale
  Baseline | 1.97 (0.82)
  Week 4 | 1.44 (0.83)
  Change at Week 4 | 0.52 (0.55)
  Week 8 | 1.02 (0.73)
  Change at Week 8 | 0.94 (0.72)
  Week 12 | 0.80 (0.70)
  Change at Week 12 | 1.14 (0.79)
  Week 16 | 0.70 (0.77)
  Change at Week 16 | 1.24 (0.91)
  Week 20 | 0.56 (0.66)
  Change at Week 20 | 1.33 (0.86)
  HAQ Week 24 | 0.56 (0.69)
  Change at Week 24 | 1.32 (0.87)

13. Secondary Outcome: Patient Global Assessment of Disease Activity (VAS)
Description: The participant's overall assessment of their current disease activity was displayed on a 100-mm horizontal VAS. The left-hand extreme (0 mm) of the line was described as "no disease activity" (symptom free and no arthritis symptoms) and the right-hand extreme (100 mm) was described as "maximum disease activity" (maximum arthritis disease activity). The change in Patient Global Assessment of Disease Activity was determined as the difference in values from baseline at each visit.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
mm
  Baseline | 64.2 (18.6)
  Week 4 | 40.6 (20.7)
  Change at Week 4 | 23.6 (21.5)
  Week 8 | 28.8 (19.8)
  Change at Week 8 | 35.6 (22.0)
  Week 12 | 21.4 (18.1)
  Change at Week 12 | 42.8 (23.8)
  Week 16 | 18.1 (19.2)
  Change at Week 16 | 46.4 (25.2)
  Week 20 | 11.3 (12.3)
  Change at Week 20 | 53.0 (22.0)
  Week 24 | 12.0 (15.3)
  Change at Week 24 | 51.6 (25.3)

14. Secondary Outcome: Physician's Global Assessment of Disease Activity (VAS)
Description: The physician's assessment of the participant's current disease activity was displayed on a 100-mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme (100 mm) was described as "maximum disease activity". The Physician's Global Assessment of Disease Activity was completed by the Efficacy Assessor who could or could not be a physician. The change in Physician's Global Assessment of Disease Activity was determined as the difference in values from baseline at each visit.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
mm
  Baseline | 61.8 (18.3)
  Week 4 | 37.7 (20.5)
  Change at Week 4 | 24.3 (20.3)
  Week 8 | 26.7 (19.4)
  Change at Week 8 | 35.4 (21.7)
  Week 12 | 20.0 (17.3)
  Change at Week 12 | 41.6 (23.5)
  Week 16 | 16.0 (18.8)
  Change at Week 16 | 46.0 (24.6)
  Week 20 | 10.0 (10.9)
  Change at Week 20 | 51.8 (21.0)
  Week 24 | 10.7 (13.2)
  Change at Week 24 | 50.6 (23.3)

15. Secondary Outcome: Patient Assessment of of Pain (VAS)
Description: The participant's assessment of their current level of pain was displayed on a 100-mm horizontal VAS. The left-hand extreme (0 mm) of the line was described as "no pain" and the right-hand extreme of the line (100 mm) was described as "unbearable pain". The change in participant's perception of pain was determined as the difference in values from baseline at each visit.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
mm
  Baseline | 63.4 (18.7)
  Week 4 | 41.4 (21.1)
  Change at Week 4 | 21.9 (20.7)
  Week 8 | 29.1 (21.0)
  Change at Week 8 | 34.5 (23.1)
  Week 12 | 21.4 (18.1)
  Change at Week 12 | 41.7 (24.1)
  Week 16 | 16.3 (17.7)
  Change at Week 16 | 46.6 (24.5)
  Week 20 | 10.6 (10.9)
  Change at Week 20 | 52.3 (21.8)
  Week 24 | 11.3 (14.3)
  Change at Week 24 | 51.5 (25.4)

16. Secondary Outcome: C-Reactive Protein (CRP)
Description: CRP is an acute phase inflammatory marker. Levels of CRP increase with inflammation. The change in CRP was determined as the difference in values from baseline and at each visit.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
mg/dL
  Baseline | 22.9 (24.1)
  Week 4 | 6.5 (14.8)
  Change at Week 4 | 16.6 (27.3)
  Week 8 | 4.9 (6.4)
  Change at Week 8 | 17.7 (23.1)
  Week 12 | 5.1 (9.4)
  Change at Week 12 | 16.8 (24.3)
  Week 16 | 5.2 (7.5)
  Change at Week 16 | 17.2 (23.3)
  Week 20 | 6.1 (11.6)
  Change at Week 20 | 16.0 (24.1)
  Week 24 | 6.7 (8.7)
  Change at Week 24 | 16.1 (24.3)

17. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR indirectly measures how much inflammation is in the body. A higher ESR is indicative of increased inflammation. The change in ESR was determined as the difference in values from baseline at each visit.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 117
mm/hr
  Baseline | 31.4 (23.3)
  Week 4 | 9.5 (11.7)
  Change at Week 4 | 21.8 (20.1)
  Week 8 | 8.3 (11.6)
  Change at Week 8 | 22.4 (20.7)
  Week 12 | 8.6 (12.0)
  Change at Week 12 | 22.9 (21.3)
  Week 16 | 8.1 (13.0)
  Change at Week 16 | 23.0 (18.9)
  Week 20 | 7.8 (11.3)
  Change at Week 20 | 22.4 (19.4)
  Week 24 | 8.2 (9.7)
  Change at Week 24 | 22.2 (2.4)

18. Primary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with adverse events (AEs), serious adverse events (SAEs), severe AEs, AEs leading to withdrawal, AEs leading to death, and treatment-related AEs.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Safety population: all participants who received at least one dose of study medication where at least one post-baseline assessment of safety was available.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 121
percentage of participants
  AEs | 48.8
  SAEs | 10.7
  With severe AEs | 8.3
  AEs leading to withdrawals | 5.8
  AEs leading to death | 0.8
  Treatment-related AEs | 10.7
  Treatment-related SAEs | 4.1
  Treatment-related severe AEs | 5.0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were recorded from the date of first infusion to the end of study visit at Week 24.
Description: An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 13/121
Other Adverse Events (participants affected / at risk) | 59/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=121)
Neutropenia (Blood and lymphatic system disorders) | 1
Hypertension (Vascular disorders) | 2
Metrorrhagia (Reproductive system and breast disorders) | 1
Hepatic cytolysis (Hepatobiliary disorders) | 3
Worsening of arthralgia (Musculoskeletal and connective tissue disorders) | 1
Necrotising fasciitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cervical cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=121)
Elevation of the AST/ALT levels (Investigations) | 22
Hypercholesterolemia (Investigations) | 18
Hypertriglyceridemia (Investigations) | 16
Bilirubin level elevations (Investigations) | 15
Neutropenia (Blood and lymphatic system disorders) | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Leucopenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 5
Increased neutrophil count (Blood and lymphatic system disorders) | 4
Joint pain (Musculoskeletal and connective tissue disorders) | 4
Hepatic cytolysis (Hepatobiliary disorders) | 4
Headache (Nervous system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Alkaline phosphatase elevations (Investigations) | 3
Bronchitis (Infections and infestations) | 3
Gingivitis (Gastrointestinal disorders) | 2
Vertigo (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Increased leukocyte count (Blood and lymphatic system disorders) | 2
Hypertension (Vascular disorders) | 2
Metrorrhagia (Reproductive system and breast disorders) | 2
Pneumonia (Infections and infestations) | 2
Oedema limbs (General disorders) | 1
Bullous lesions (Skin and subcutaneous tissue disorders) | 1
Necrotising fasciitis (Infections and infestations) | 1
Stiffness (Musculoskeletal and connective tissue disorders) | 1
Fever (General disorders) | 1
Gastralgia (Gastrointestinal disorders) | 1
Swelling of the upper and lower limbs (General disorders) | 1
Chest pain (General disorders) | 1
Tooth abscess (Infections and infestations) | 1
Zona (General disorders) | 1
Inguinal adenopathy (Blood and lymphatic system disorders) | 1
Inflammation at the site of infusion (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Tingling (Nervous system disorders) | 1
Chills (General disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Decreased level of HDL cholesterol (Investigations) | 1
Elevation of creatine level (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.